CLINICAL TRIAL: NCT07212426
Title: A Phase II, Multicenter, Randomized, Open-Label Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of LP-005 Injection in Patients With Paroxysmal Nocturnal Hemoglobinuria.
Brief Title: Efficacy, Safety, and Pharmacokinetics of LP-005 Injection in PNH Patients.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Longbio Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P10-LP005-02
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: PNH - Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LP-005 900 mg (Experimental): Patients will receive intravenous infusion of LP-005 Injection at a dose of 900 mg once every 4 weeks.
  Interventions: Biological: LP-005 Injection
- LP-005 1200 mg (Experimental): Patients will receive intravenous infusion of LP-005 Injection at a dose of 1200 mg once every 4 weeks.
  Interventions: Biological: LP-005 Injection
- LP-005 1500 mg (Experimental): Patients will receive intravenous infusion of LP-005 Injection at a dose of 1500 mg once every 4 weeks.
  Interventions: Biological: LP-005 Injection

INTERVENTIONS:
Biological: LP-005 Injection — IV infusion, Q4W

SUMMARY:
This is a multicenter, randomized, open-label, Phase II clinical study to evaluate the efficacy, safety, and pharmacokinetics of LP-005 injection in adult patients with paroxysmal nocturnal hemoglobinuria (PNH).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 years.
* Diagnosis of PNH based on flow cytometry with clone size > 10% by granulocytes.
* Presence of one or more PNH-related signs or symptoms within 3 months prior to screening or a history of transfusion due to PNH.
* LDH level ≥2.0×upper limit of the normal range(ULN).
* Hemoglobin level <100 g/L at screening.

Exclusion Criteria:

* Active or suspected active viral, bacterial, fungal, or parasitic infection within 14 days prior to screening.
* History of meningococcal infection.
* History of splenectomy or congenital asplenia.
* History of systemic autoimmune disease or known/suspected immunodeficiency.
* History of hematopoietic stem cell transplantation.
* Use of any complement inhibitor within 3 months prior to screening or within 5 drug half-lives (whichever is longer).
* Pregnant or breastfeeding women, or women planning to become pregnant during the study or follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-14 (Actual); Primary Completion 2026-05-06 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in serum lactate dehydrogenase (LDH) levels. | Baseline and at Week 12.
Proportion of participants with ≥2 g/dL increase in hemoglobin level from Baseline in the absence of transfusion. | Baseline and at Week 24.

SECONDARY OUTCOMES:
Proportion of participants with ≥2 g/dL increase in hemoglobin level from Baseline in the absence of transfusion. | Baseline and at Week 12 and 48
Proportion of participants who are transfusion-free. | Baseline to Week 12, 24 and 48
Change from Baseline in the number of red blood cell (RBC) transfusions. | Baseline to Week 24 and 48.
Change from Baseline in hemoglobin levels. | Baseline, Week 12, 24 and 48
Proportion of participants achieving hemoglobin levels ≥100 g/L in the absence of transfusion. | Baseline, Week 12, 24 and 48
Proportion of participants with LDH levels normalized. | Baseline, Week 12, 24 and 48
Changes in serum complement hemolytic activity. | Observation from Predose on Day 1 through 337 days post-administration.
Change From Baseline in Fatigue as Measured by Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Baseline and at Week 12, 36, and 48.
  FACIT-F is a 40-item measure that assesses self-reported fatigue and its impact upon daily activities and function. The higher the score, the better the QOL.
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs). | Baseline up to approximately 13 months.
Serum concentrations of LP-005. | Observation from Predose on Day 1 through 337 days post-administration.
Number of Participants with Treatment-emergent Anti-Drug Antibodies (ADA) and neutralizing antibodies (Nab) Response to LP-005. | Observation from Predose on Day 1 through 337 days post-administration.

CONTACTS AND LOCATIONS:
Overall Officials: Guangsheng He, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China